CLINICAL TRIAL: NCT02990221
Title: A Randomized Study to Evaluate the Efficacy of Ingenol Mebutate on Actinic Keratoses and Field Cancerization Compared to Cryotherapy
Brief Title: Efficacy of Ingenol Mebutate on Actinic Keratoses and Field Cancerization vs Cryotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Giuseppe Argenziano, Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIS-PICATO 1264
Record Dates: First submitted 2016-12-02; First posted 2016-12-13 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Actinic Keratosis
Keywords: Field Cancerization
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate; Cryotherapy; Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ingenol mebutate (Active Comparator): application of ingenol mebutate for 3 consecutive days on an area of face/scalp of 25 cm2
  Interventions: Drug: Ingenol mebutate
- cryotherapy (Active Comparator): application of criotherapy on actinic keratosis present in an area of face/scalp of 25 cm2 different from the ingenol mebutate area
  Interventions: Procedure: cryotherapy

INTERVENTIONS:
Drug: Ingenol mebutate — 150 mcg / g per day, to be applied on a predetermined area of 25 cm2 of skin of the face or scalp, for 3 days consecutive
  Other Names: Picato
  Arms: Ingenol mebutate
Procedure: cryotherapy — application with 5 seconds of freezing time of each lesion located in a predetermined skin area of 25 cm2 of the face or scalp
  Other Names: cryosurgery
  Arms: cryotherapy

SUMMARY:
The main objective of this study is to compare the effectiveness of ingenol mebutate gel (150 mcg / g per day, to be applied on a predetermined area of 25 cm2 of skin of the face or scalp, for 3 days consecutive) cryotherapy (application with 5 seconds of freezing time of each lesion located in a predetermined skin area of 25 cm2 of the face or scalp) in the treatment of actinic keratosis and their field cancerization.

Study details:

This study is randomized. 50 subjects with at least two actinic keratoses of grade I and II, located in two different districts of 25 cm2 skin of the face or scalp, and who meet all the inclusion criteria will be enrolled in the study by the investigators in the three different centers mentioned above.

The investigators will assess the effect of treatment by confocal microscopy and digital dermoscopy. The investigator will acquire images of selected areas of the face and scalp before and after treatment. Data will be collected and analyzed by the coordinating centre.

Procedure for the study:

Recruitment of subjects; random assignment of treatment (ingenol mebutate gel 150 micrograms/g and cryotherapy) to the two skin areas of 25 cm2 of the subject recruited; evaluation of the two areas with reflectance confocal microscopy and digital dermoscope. The measurements will be carried out at time 0, after 1 month and 6 months. The investigator must fill out a form for each subject at the beginning (day 0), after 1 month and at the end of the study (after 6 months). The subject must complete a questionnaire at the beginning (day 0), after 1 month and at the last follow-up visit (after 6 months).

Measurement parameters: Dermoscopy and confocal microscopy will be used to assess the percentage reduction in actinic keratoses and the damage of the cancerous area in the two selected areas treated with ingenol mebutate gel or cryotherapy, respectively.

Adverse / side events will be collected at each visit by the investigator and will be contained in another form.

DETAILED DESCRIPTION:
This study is designed to compare the efficacy of topical ingenol mebutate (150 mcg/g once daily on a selected facial or scalp target area of 25 cm2, for 3 consecutive days) with cryosurgery (applied for a freeze time of 5 seconds, on each lesion included in an area of 25 cm2 on face or scalp)

This is a national, post-marketing (phase 4), on label, interventional, randomized trial.

Subjects will attend a screening visit where they will be assessed for eligibility.

Two areas of treatment in the same patient have to be identified (e.g. scalp and cheek or two different part of the balding scalp), than these two areas will be randomized in a 2:1 ratio: one will be treated with cryosurgery and the other one with Picato Gel.

The cryosurgery will be performed in the same day during the visit (1 application for a freeze time of 5 seconds, on each lesion included in an area of 25 cm2 on face or scalp) Picato gel 150 mcg will be applied at home by the patient, according to current indication (RCP: 3 consecutive days for a total of three application in an area of 25 cm2) Subjects will be followed for 24 weeks (about 6 months) after the cryosurgery application (Visit 1).

Adverse events and patient compliance will be recorded 7 days after cryosurgery application and 5 days after first Picato gel application (Visit 2). The number of AKs present within the treatment areas will be counted at Visit 1 (Baseline AK count) and at Visits 3 - 4 (AKcount). The data obtained will provide information on the effect of Picato gel versus Cryosurgery on recurrence rate of AKs.

Furthermore, the trial will also provide data on the effect of Picato gel versus Cryosurgery on the appearance rate of new AKs.

The final results for all subjects will be included in a Final Clinical Study Report in the original submission. This includes final results for all primary and secondary endpoints as well as 6-month recurrence and Adverse Event data.

ELIGIBILITY:
Inclusion Criteria:

A patient will be enrolled if he/she meets all of the following inclusion criteria:

* Current diagnosis of AK, with ≥2 lesions of grade I and/or II located in two different anatomical districts (within a contiguous 25 cm2 area on the face, scalp or forehead);
* Male ≥ 18 years of age or Female > 60 years of age;
* Skin type I or II according to Fitzpatrick;
* Patient has confirmed his/her willingness to participate in this study after being informed of all aspects of the study that are relevant to his/her decision to participate, by signing and dating the approved informed consent form, according to ICH and local laws.

The 25 cm2 contiguous treatment areas could be of any shape, e.g. 5 cm x 5 cm, 2 cm x 12.5 cm, 3 cm x 8.3 cm.

Exclusion Criteria:

A patient will be excluded if he/she meets any of the following exclusion criteria:

* Has received any therapy for AK within the past 3 months
* Has AK of grade III
* Has currently a skin cancer or shows an early stage of skin cancer;
* Has another skin disease that requires treatment with other medications in the AK area or in distance of 3 cm;
* Use of cosmetic or therapeutic products and procedures which could interfere with assessments of the treatment area;
* Immunosuppressive therapies or current treatment for cancer;
* Clinically unstable medical condition;
* High risk group for HIV infection or presentation of other infectious diseases (hepatitis A virus , hepatitis B virus , hepatitis C virus , Tuberculosis, etc);
* Allergies to the tested gel (ingenol mebutate and eccipients);
* Pregnancy and breastfeeding (see inclusion criteria);
* Psychiatric disease that may interfere with follow-up of study procedures;
* Participation in other clinical trials up to 30 days prior to day 1 of the study;
* Patient is, for any reason, considered by the investigator to be an unsuitable candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
At least 75% reduction in the total AK count relative to baseline | 6-month follow-up
  The primary efficacy endpoint is the percentage change, at the end of the treatment period, in the number of AK lesions that were originally defined in the selected AK target area at baseline. The percentage change in the number of AK lesions is calculated as the number of lesions present at the end of the treatment period in the target area minus the number of AK lesions present in the target area at baseline visit divided by the number of lesions present in the target area at baseline. This variable will be analysed using a non-parametric analysis (Wilcoxon Rank-sum test).
Reduction of subclinical AK lesions according to a Reflectance Confocal Microscopy score | 6-month follow-up
  Change from baseline in RCM score of target area and RCM score of cancerization field at the end of the treatment period. Each of the 13 RCM criteria will be scored 0 (absent), 1 (<25%), 2 (25%-50%), 3 (50-75%), or 4(>75%). An overall score will be obtained by averaging the RCM scores at the epidermal, DEJ and dermal level. The same approach will be used for the RCM examination of the cancerization field. The above variables will be compared between the groups using a t-test, 95% confidence interval for the between-group difference will be provided.

SECONDARY OUTCOMES:
Absence of new lesions after a follow-up period of 6 months | 6-month follow-up
  The count of AK lesions will be performed by exploration and palpation (numeric count) and the presence will be also confirmed by dermoscopic assessment (numeric count)
cosmetic outcome | 6-month follow-up
  cosmetic outcome will be evaluated by Patient's assessment of satisfaction to product at the end of the treatment period (specific questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Argenziano, Prof, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Second University of Naples, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Frost CA, Green AC. Epidemiology of solar keratoses. Br J Dermatol. 1994 Oct;131(4):455-64. doi: 10.1111/j.1365-2133.1994.tb08544.x. PMID 7947197
- [Result] Fu W, Cockerell CJ. The actinic (solar) keratosis: a 21st-century perspective. Arch Dermatol. 2003 Jan;139(1):66-70. doi: 10.1001/archderm.139.1.66. No abstract available. PMID 12533168
- [Result] Ortonne JP. From actinic keratosis to squamous cell carcinoma. Br J Dermatol. 2002 Apr;146 Suppl 61:20-3. doi: 10.1046/j.1365-2133.146.s61.6.x. PMID 11966728
- [Result] Cohen JL. Actinic keratosis treatment as a key component of preventive strategies for nonmelanoma skin cancer. J Clin Aesthet Dermatol. 2010 Jun;3(6):39-44. PMID 20725550
- [Result] Padilla RS, Sebastian S, Jiang Z, Nindl I, Larson R. Gene expression patterns of normal human skin, actinic keratosis, and squamous cell carcinoma: a spectrum of disease progression. Arch Dermatol. 2010 Mar;146(3):288-93. doi: 10.1001/archdermatol.2009.378. PMID 20231500
- [Result] Vatve M, Ortonne JP, Birch-Machin MA, Gupta G. Management of field change in actinic keratosis. Br J Dermatol. 2007 Dec;157 Suppl 2:21-4. doi: 10.1111/j.1365-2133.2007.08268.x. PMID 18067627
- [Result] Fidler B, Goldberg T. Ingenol mebutate gel (picato): a novel agent for the treatment of actinic keratoses. P T. 2014 Jan;39(1):40-6. PMID 24672213
- [Result] Andrews MD. Cryosurgery for common skin conditions. Am Fam Physician. 2004 May 15;69(10):2365-72. PMID 15168956